CLINICAL TRIAL: NCT01402232
Title: REduction of rIsk for Contrast-Induced Nephropathy (REICIN) Study:RESCIND-P (Prospective Observational Study for REduction of contraSt-induced Nephropathy and Cardiaovascular Events followINg carDiac Catheterization)
Brief Title: REduction of rIsk for Contrast Induced Nephropathy
Acronym: REICIN-RESCIND
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Nanfang Hospital, Southern Medical University (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Guangdong Medical College (Other); Dongguan Kanghua Hospital (Other); Dongguan People's Hospital (Other Government); Maoming People's Hospital (Other); Futian People's Hospital (Other); Longyan City First Hospital (Other); First People's Hospital of Kashgar (Unknown)
Responsible Party: Principal Investigator, Jiyan Chen, MD, Guangdong Provincial People's Hospital
Other Study IDs: Y20110721
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Contrast Induced Nephropathy
Keywords: contrast-induced nephropathy; contrast medium; creatinine clearance; coronary angiography; diabetes; chronic kidney disease; predictive
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- coronary angiography: We recruit all consecutive patients who were undergoing coronary angiography or percutaneous coronary intervention.

SUMMARY:
The REduction of rIsk for Contrast-Induced Nephropathy (REICIN) study is the largest prospective multicenter data base for CIN flowing coronary angiography (CAG) or percutaneous coronary intervention (PCI). The REICIN study has the potential to characterize contemporary CIN incidence, modified risk factors and prognosis, so that to identify strategiaes to reduce risk of CIN following CAG/PCI.

DETAILED DESCRIPTION:
This is a multicenter prospective observational study collecting data on over 5000 CAG patients admitted to department of cardiology in 12 hospitals from January 2013. Data will be collected for more than 1 year on all patients undergoing CAG with or without PCI older than 18 years without baseline end-stage renal failure needing renal replacement therapy or renal transplantation. Data to be collected includes demographic information, admission diagnoses and co-morbidities, biomarkers and details on preventive hydration and medications used Contrast-induced nephropathy (CIN) is the primary endpoint, defined as a ≥ 0.5 mg/dL or 25% increase in serum creatinine (SCr) from baseline during the first 48 to 72 hours after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred to CAG or PCI;
2. Age ≥ 18 years
3. Submit informed consent and adhere to the study protocol

Exclusion Criteria:

1. Fail to undergo CAG/PCI or die during the procedure；
2. End-stage renal diseases or renal replacement；
3. Pre-procedural unstable renal funciton (acute increase in serum creatinine more than 0.5mg/ml in the past 24 h)；
4. Intravascular administration of a contrast medium within the previous 48 hours；
5. Allergic to contrast medium;
6. Pregnancy, lactation or malignant tumoror life expectancy< 1 year;
7. The use of renal toxicity drugs (non-steroidal anti-inflammatory drugs, aminoglycoside drugs, cyclosporine, cisplatin etc) within 48 h before cardiac catheter surgery and the whole process of the research;
8. Refer to receive renal artery angiography or surgical valve replacement in patients with rheumatic heart disease； For exclusion creteria 7, patients admited and taked aspirin are included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We reviewed all consecutive patients who were undergoing coronary angiography
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-02 (Actual); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
contrast-induced nephropathy | 48-72 h
  Contrast-Induced Nephropathy was defined as a ≥ 0.5 mg/dL or 25% increase in serum creatinine from baseline during the first 48 to 72 hours after the procedure.

SECONDARY OUTCOMES:
contrast-induced acute kidney injury (CI-AKI0.3) | 48h
  defined as a ≥ 0.3 mg/dL absolute increase in serum creatinine from baseline during the first 48 hours after the procedure
Cystatin C based CI-AKI (CI-AKIcyc) | 24-48h
  defined as a ≥10% absolute increase in serum cystatin C during the first 24 hours after the procedure and and a ≥ 0.3 mg/dL absolute increase in serum creatinine from baseline during the first 48 hours after the procedure.
The change of eGFR, calculate based on CrCl and serum cystatin C | 48-72 h
  The eGFRcreatinine-cystatin C was calculated by the 2012 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) cystatin C equation: 135 × min(Scr/κ, 1)α × max(Scr/κ, 1)-0.601 × min(Scys/0.8, 1)-0.375 × max (Scys/0.8, 1)-0.711 × 0.995Age [× 0.969 if female] [× 1.08 if black], where Scr is serum creatinine, Scys is serum cystatin C, κ is 0.7 for females and 0.9 for males, α is -0.248 for females and -0.207 for males, min indicates the minimum of Scr/κ or 1, and max indicates the maximum of Scr/κ or 1.
Persistent CI-AKI (CI-AKIp) | 3 months
  defined as residual impairment of renal function indicated by a ≥ 25% reduction in creatinine clearance at 3 months in comparison with baseline.
In-hospital major adverse cardiovascular and clinical events | In-hospital
  all-cause mortality (cardiovascular and noncardiovascular), required renal replacement therapy (RRT), cardiovascular events (acute myocardial infarction, acute heart failure，cardiac shock, heart/ventricular septal rupture,clinical arrhythmia), Cerebrovascular events (Stroke), and bleeding (TIMI grade) .
Follow-up major adverse cardiovascular and clinical events | >=1 year
  all-cause mortality, RRT, re-hospitalization, cardiovascular events, cerebrovascular events, and bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Liu, MD,PhD, Study Director — Guangdong Cardiovascular Institute,Guangdong General Hospital; Shiqun Chen, MS, Study Director — Guangdong Cardiovascular Institute,Guangdong General Hospital
Locations (12):
- China (12):
  - Kaihong Chen, Longyan, Fujian
  - Guoliang Jia, Dongguan, Guangdong
  - Jianfeng Ye, Dongguan, Guangdong
  - Jian Qiu, Guangzhou, Guangdong
  - Jingfeng Wang, Guangzhou, Guangdong
  - Ken Wu, Guangzhou, Guangdong
  - Yuqing Hou, Guangzhou, Guangdong
  - Zhiming Du, Guangzhou, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Yan Liang, Maoming, Guangdong
  - Guifu Wu, Shenzhen, Guangdong
  - Xiaoguang Zhou, Kashgar, Xinjiang